CLINICAL TRIAL: NCT03746184
Title: The Right Treatment for the Right Patient At the Right Time - a Prospective Cohort Study of 5,000 Patients with Knee Osteoarthritis
Brief Title: The Right Treatment for the Right Patient At the Right Time. a Study Following 5,000 Patients with Knee Osteoarthritis
Acronym: TREATright
Status: Active, not recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Naestved Hospital (Other); University of Copenhagen (Other); VIVE - The Danish Center for Social Science Research (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anders Troelsen, Professor, consultant, dr.med., PhD, Hvidovre University Hospital
Other Study IDs: CAGROAD_TREATright_2018
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: precision medicine; Patient-Specific Modeling
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Knee osteoarthritis: Treatment course
  Interventions: Other: Treatment course

INTERVENTIONS:
Other: Treatment course — Pursued treatment for knee OA, including type of health care provider, time period of treatment course, and types of treatments received, will be recorded via the patient-reported questionnaire.

SUMMARY:
The treatment that patients with knee OA are offered varies largely. There is a need for more evidence-based individualized guidance to treatment choice for knee osteoarthritis. This study will register and evaluate the course and outcome of treatment in 5,000 patients with knee osteoarthritis. The understanding of knee OA treatment will advance in three ways: Firstly, by describing the different treatment pathways that are currently being used for knee OA. Secondly, by identifying wich individual factors that may impact the outcome of the treatment course. And finally, by conducting the economic burden related to different treatment modalities.

DETAILED DESCRIPTION:
The problem: Knee Osteoarthritis (OA), the most common form of arthritis, is a chronic, widespread disease with a steadily increasing prevalence that places a major economic burden on the society. Patients with knee OA suffer from chronic knee pain and functional disabilities. The treatment that patients with knee OA are offered varies largely, and is often not in coherence with clinical guidelines. The guidelines recommend patient education, exercise, and weight control as core interventions for all patients with knee OA and surgical intervention for end-stage knee OA. However, the timing of surgery is debated, and whether the outcome of different treatment strategies depend on individual factors such as the patients symptoms, OA severity, or prior treatment, has not been established.

The solution: This large-scale study aims at improving the understanding of which treatment should be offered to which patient with knee OA at which time. The study is an interdisciplinary, collaborative effort, including orthopaedic surgeons, physiotherapists and general practitioners from two different regions in Denmark. At least 5,000 patients with primary referrals to orthopaedic surgeons due to knee OA, at two public hospitals, will be recruited through a two-year inclusion period. Patients' prior treatment and symptom severity will be registered at the first consultation with the orthopaedic surgeon using a patient self-reported questionnaire. OA severity will be defined on plain standing knee radiographs using a well-established classification system. The course of treatment will be registered after 6 months and 2 years through a self-reported questionnaire with additional questions asking whether patients can accept their current symptom state, or, if not, whether they consider the treatment to have failed.

Societal impact and clinical implications: The understanding of knee OA treatment will advance in three ways: Firstly, our results will improve the overview by describing the different treatment pathways that are currently being used for knee OA. Secondly, predictors of good and poor treatment outcomes of different treatment modalities, or combinations hereof will be identified. And finally, the cost-effectiveness of different treatment modalities will be evaluated. These results will be used to develop a treatment algorithm to help patients with knee OA and clinicians to tailor the right treatment at the right time through shared decision-making.

ELIGIBILITY:
Inclusion Criteria:

* primary referrals to one of two orthopedic department's outpatient clinics due to knee osteoarthritis

Exclusion Criteria:

* previous total or unicompartmental knee replacement
* osteotomy around the study knee
* unable to read or write Danish
* patients who decline to answer the questionnaire at inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with primary referrals to one of two public hospitals orthopedic department's outpatient clinics due to knee osteoarthritis are consecutively invited to participate. The two hospitals cover the larger part of Zealand in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Acceptable Symptom State (PASS) | 2 years after inclusion
  Patients answer yes/no to a PASS question asking whether they consider the current symptom state to be acceptable.
Treatment Failure | 2 years after inclusion
  Patients who answer "no" to the PASS question will also answer "yes/no" to a question about whether they consider the treatment received to have failed.

SECONDARY OUTCOMES:
Patient Acceptable Symptom State (PASS) | 6 months after inclusion
  Patients answer yes/no to a PASS question asking whether they consider the current symptom state to be acceptable.
Treatment Failure | 6 months after inclusion
  Patients who answer "no" to the PASS question will also answer "yes/no" to a question about whether they consider the treatment received to have failed.
Minimal Important Change | 6 months and 2 years after inclusion
  An anchor question asking about the degree and importance of change in knee-pain and function will be answered on a 7-level Likert scale ranging from better, an important improvement to worse, an important deterioration.
Oxford Knee Score (OKS), range from 0 (worst) to 48 (best) | 6 months and 2 years after inclusion
  Patient self-reported average knee pain and function during the past four weeks calculated from a validated 12-item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, Professor, Study Chair — Copenhagen University Hospital, Hvidovre; Lina H Ingelsrud, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Henrik M Schroeder, Asst. Prof., Study Chair — Næstved Sygehus, Denmark; Søren T Skou, Assoc. Prof., Study Chair — Næstved-Slagelse-Ringsted Hospitals AND University of Southern Denmark; Thomas Bandholm, Professor, Study Chair — University of Copenhagen AND Copenhagen University Hospital Hvidovre, Denmark; Jakob Kjellberg, Professor, Study Chair — VIVE - The Danish Centre of Applied Social Science, Denmark; Susanne Reventlow, Professor, Study Chair — University of Copenhagen; Anne Møller, Asst. Prof., Study Chair — University of Copenhagen; Simon M Bruhn, M.Sc., Study Chair — Copenhagen University Hospital, Hvidovre
Locations (1):
- Department of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Decision in pending on whether the total database with all anonymised data will be transferred to the Danish National Archives' Collections once the study is completed.

REFERENCES:
- [Derived] Bruhn SM, Skou ST, Harris LK, Bandholm T, Moller A, Schroder HM, Troelsen A, Ingelsrud LH. Usage of guideline-adherent core treatments for knee osteoarthritis before and after consulting an orthopaedic surgeon: A prospective cohort study. Osteoarthr Cartil Open. 2023 Sep 28;5(4):100411. doi: 10.1016/j.ocarto.2023.100411. eCollection 2023 Dec. PMID 37818279
- [Derived] Bruhn SM, Ingelsrud LH, Bandholm T, Skou ST, Schroder HM, Reventlow S, Moller A, Kjellberg J, Kallemose T, Troelsen A. Disentangling treatment pathways for knee osteoarthritis: a study protocol for the TREATright study including a prospective cohort study, a qualitative study and a cost-effectiveness study. BMJ Open. 2021 Jul 7;11(7):e048411. doi: 10.1136/bmjopen-2020-048411. PMID 34233992